CLINICAL TRIAL: NCT04270370
Title: A Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of Single-and Multiple Ascending Doses of LY3478045in Healthy Subjects
Brief Title: A Study of LY3478045 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17537; J2M-MC-GZKA (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3478045 (Part A) (Experimental): Participants received single ascending oral dose of 20 milligram (mg), 60mg, 180 mg, 500 mg, 700 mg LY3478045 on Day 1.
  Interventions: Drug: LY3478045
- Placebo (Part A) (Placebo Comparator): Participants received single oral dose of placebo on Day 1.
  Interventions: Drug: Placebo
- LY3478045 (Part B) (Experimental): Participants received multiple ascending oral dose of 60mg and 300 mg LY3478045 once-daily (QD)for 14 days.
  Interventions: Drug: LY3478045
- Placebo (Part B) (Placebo Comparator): Participants received oral dose of placebo QD for 14 days.
  Interventions: Drug: Placebo
- LY3478045 + Atorvastatin (Part B) (Experimental): Participants received multiple ascending oral doses of 160 mg, 360 mg LY3478045 QD for 14 days and 40 mg atorvastatin administered orally 4 hours after breakfast on Day -2 and 4 hours after LY3478045 administration on Day 7.
  Interventions: Drug: LY3478045; Drug: Atorvastatin
- Placebo + Atorvastatin (Part B) (Placebo Comparator): Participants received oral dose of placebo QD for 14 days and 40 mg atorvastatin administered orally 4 hours after breakfast on Day -2 and 4 hours after LY3478045 administration on Day 7.
  Interventions: Drug: Placebo; Drug: Atorvastatin

INTERVENTIONS:
Drug: LY3478045 — Administered orally.
  Arms: LY3478045 (Part A); LY3478045 (Part B); LY3478045 + Atorvastatin (Part B)
Drug: Placebo — Administered orally.
  Arms: Placebo (Part A); Placebo (Part B); Placebo + Atorvastatin (Part B)
Drug: Atorvastatin — Administered orally.
  Arms: LY3478045 + Atorvastatin (Part B); Placebo + Atorvastatin (Part B)

SUMMARY:
The main purpose of this study in healthy participants is to learn more about the safety of LY3478045 and any side effects that might be associated with it. The study will also measure how much LY3478045 gets into the bloodstream and how long it takes the body to get rid of it.

This study has two parts: Part A (one dose) will last about six weeks and Part B (more than one dose) will last about eight weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy participants as determined through medical history and physical examination
* Have a body mass index greater than or equal to (≥)18.5 and less than or equal to (≤)40 kilograms per square meter (kg/m²)
* Have had a stable weight for 3 months prior to screening and enrollment (less than [<]5 percent [%] body weight change) and have not received dietary intervention in the 3 months prior to screening and enrollment
* Have safety laboratory test results within the normal reference range for the population or investigative site, or results with acceptable deviations that are judged as not clinically significant by the investigator

Exclusion Criteria:

* Have a history of fructosuria
* Have an abnormality in the 12-lead electrocardiogram (ECG) at screening that, in the opinion of the investigator, increases the risks associated with participating in the study or may confound ECG (QT) data analysis
* Have blood pressure greater than (>)160/90 millimeters of mercury (mmHg) and pulse rate <50 or >100 beats per minute (bpm), supine (at screening), or with minor deviations judged to be acceptable by the investigator
* Use of any drugs or substances that are known strong inducers or inhibitors of cytochrome P450 (CYP)3A or organic anion-transporting polypeptides (OATPs) are specifically excluded within 14 days prior to the first administration of study drug and during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included two parts (Part A and Part B). A single ascending oral dose of LY3478045 was administered in Part A, and multiple ascending oral doses of LY3478045 were administered once daily (QD) in Part B. Participants in a few reporting arms of Part B received a 40-milligram (mg) oral dose of atorvastatin 4 hours after breakfast on Day -2 and 4 hours after LY3478045 administration on Day 7.
Groups:
- 20 mg LY3478045 (Part A): Participants received single oral dose of 20 mg LY3478045 on Day 1.
- 60 mg LY3478045 (Part A): Participants received single oral dose of 60 mg LY3478045 on Day 1.
- 180 mg LY3478045 (Part A): Participants received single oral dose of 180 mg LY3478045 on Day 1.
- 500 mg LY3478045 (Part A): Participants received single oral dose of 500 mg LY3478045 on Day 1.
- 700 mg LY3478045 (Part A): Participants received single oral dose of 700 mg LY3478045 on Day 1.
- Placebo Once-daily (QD) (Part B): Participants received oral dose of Placebo QD for 14 days.
- Placebo QD + 40 mg Atorvastatin (Part B): Participants received oral dose of placebo QD for 14 days and 40 mg atorvastatin administered orally 4 hours after breakfast on Day -2 and 4 hours after LY3478045 administration on Day 7.
- 60 mg LY3478045 QD (Part B): Participants received oral dose of 60 mg LY3478045 QD for 14 days.
- 160 mg LY3478045 QD + 40 mg Atorvastatin (Part B): Participants received oral dose of 160 mg LY3478045 QD for 14 days and 40 mg atorvastatin administered orally 4 hours after breakfast on Day -2 and 4 hours after LY3478045 administration on Day 7.
- 300 mg LY3478045 QD (Part B): Participants received oral dose of 300 mg LY3478045 QD for 14 days.
- 360 mg LY3478045 QD + 40 mg Atorvastatin (Part B): Participants received oral dose of 360 mg LY3478045 for 14 days and 40 mg atorvastatin administered orally 4 hours after breakfast on Day -2 and 4 hours after LY3478045 administration on Day 7.
Period: Overall Study
Arm/Group | Placebo (Part A) | 20 mg LY3478045 (Part A) | 60 mg LY3478045 (Part A) | 180 mg LY3478045 (Part A) | 500 mg LY3478045 (Part A) | 700 mg LY3478045 (Part A) | Placebo Once-daily (QD) (Part B) | Placebo QD + 40 mg Atorvastatin (Part B) | 60 mg LY3478045 QD (Part B) | 160 mg LY3478045 QD + 40 mg Atorvastatin (Part B) | 300 mg LY3478045 QD (Part B) | 360 mg LY3478045 QD + 40 mg Atorvastatin (Part B)
Started | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6 | 6 | 6
Received at Least One Dose of Study Drug | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6 | 6 | 6
Completed | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 5 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Placebo QD (Part B): Participants received oral dose of placebo QD for 14 days.
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | 20 mg LY3478045 (Part A) | 60 mg LY3478045 (Part A) | 180 mg LY3478045 (Part A) | 500 mg LY3478045 (Part A) | 700 mg LY3478045 (Part A) | Placebo QD (Part B) | Placebo QD + 40 mg Atorvastatin (Part B) | 60 mg LY3478045 QD (Part B) | 160 mg LY3478045 QD + 40 mg Atorvastatin (Part B) | 300 mg LY3478045 QD (Part B) | 360 mg LY3478045 QD + 40 mg Atorvastatin (Part B) | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6 | 6 | 6 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (9.4) | 43.0 (12.0) | 40.2 (13.7) | 42.3 (9.1) | 47.8 (7.6) | 50.5 (9.6) | 52.0 (4.7) | 48.3 (7.5) | 35.8 (12.8) | 36.5 (9.9) | 48.0 (9.6) | 54.8 (6.4) | 44.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 3 | 3 | 3 | 3 | 2 | 2 | 0 | 6 | 6 | 35
  Male | 6 | 5 | 4 | 3 | 3 | 3 | 1 | 2 | 4 | 6 | 0 | 0 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 1 | 3 | 3 | 3 | 1 | 1 | 2 | 1 | 3 | 2 | 27
  Not Hispanic or Latino | 6 | 3 | 5 | 3 | 3 | 3 | 3 | 3 | 4 | 5 | 3 | 4 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 3 | 3 | 2 | 1 | 2 | 2 | 2 | 2 | 4 | 4 | 3 | 1 | 29
  White | 7 | 3 | 4 | 5 | 4 | 4 | 2 | 2 | 2 | 1 | 3 | 5 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6 | 6 | 6 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, is reported in the Reported Adverse Events module.
Time Frame: Baseline Up to Final Follow-up: Up to 14 Days (Part A) and up to 28 Days (Part B)
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo (Part A) | 20 mg LY3478045 (Part A) | 60 mg LY3478045 (Part A) | 180 mg LY3478045 (Part A) | 500 mg LY3478045 (Part A) | 700 mg LY3478045 (Part A) | Placebo QD (Part B) | Placebo QD + 40 mg Atorvastatin (Part B) | 60 mg LY3478045 QD (Part B) | 160 mg LY3478045 QD + 40 mg Atorvastatin (Part B) | 300 mg LY3478045 QD (Part B) | 360 mg LY3478045 QD + 40 mg Atorvastatin (Part B)
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of LY3478045
Description: PK: AUC(0-inf) of LY3478045 was reported.
Time Frame: Part A: Predose, 0.75, 1.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72 and 95 hours post dose; Part B: Day 1: Predose, 0.75, 1.5, 3, 4, 6, 8, 12, 16 and 24 hours post dose; Day 14: Predose ,0.75, 1.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/ mL)
Arm/Group | 20 mg LY3478045 (Part A) | 60 mg LY3478045 (Part A) | 180 mg LY3478045 (Part A) | 500 mg LY3478045 (Part A) | 700 mg LY3478045 (Part A) | 60 mg LY3478045 QD (Part B) | 160 mg LY3478045 QD + 40 mg Atorvastatin (Part B) | 300 mg LY3478045 QD (Part B) | 360 mg LY3478045 QD + 40 mg Atorvastatin (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*h/ mL) | 7410 (38) | 24300 (51) | 59900 (32) | 275000 (39) | 382000 (19) | 67800 (154) | 98900 (37) | 388000 (71) | 484000 (48)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) of LY3478045
Description: PK: Cmax of LY3478045 was reported.
Time Frame: as for outcome 2
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 20 mg LY3478045 (Part A) | 60 mg LY3478045 (Part A) | 180 mg LY3478045 (Part A) | 500 mg LY3478045 (Part A) | 700 mg LY3478045 (Part A) | 60 mg LY3478045 QD (Part B) | 160 mg LY3478045 QD + 40 mg Atorvastatin (Part B) | 300 mg LY3478045 QD (Part B) | 360 mg LY3478045 QD + 40 mg Atorvastatin (Part B)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 303 (25) | 1280 (34) | 3670 (24) | 14500 (28) | 18500 (34) | 2360 (40) | 5920 (33) | 19500 (19) | 22400 (27)

ADVERSE EVENTS:
Time Frame: Baseline Up to Final Follow-up: Up to 14 Days (Part A) and up to 28 Days (Part B)
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | Placebo (Part A) | 20 mg LY3478045 (Part A) | 60 mg LY3478045 (Part A) | 180 mg LY3478045 (Part A) | 500 mg LY3478045 (Part A) | 700 mg LY3478045 (Part A) | Placebo QD (Part B) | Placebo QD + 40 mg Atorvastatin (Part B) | 60 mg LY3478045 QD (Part B) | 160 mg LY3478045 QD + 40 mg Atorvastatin (Part B) | 300 mg LY3478045 QD (Part B) | 360 mg LY3478045 QD + 40 mg Atorvastatin (Part B)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 2/10 | 1/6 | 0/6 | 2/6 | 1/6 | 1/6 | 1/4 | 2/4 | 0/6 | 0/6 | 1/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=10) | 20 mg LY3478045 (Part A) (N=6) | 60 mg LY3478045 (Part A) (N=6) | 180 mg LY3478045 (Part A) (N=6) | 500 mg LY3478045 (Part A) (N=6) | 700 mg LY3478045 (Part A) (N=6) | Placebo QD (Part B) (N=4) | Placebo QD + 40 mg Atorvastatin (Part B) (N=4) | 60 mg LY3478045 QD (Part B) (N=6) | 160 mg LY3478045 QD + 40 mg Atorvastatin (Part B) (N=6) | 300 mg LY3478045 QD (Part B) (N=6) | 360 mg LY3478045 QD + 40 mg Atorvastatin (Part B) (N=6)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=10) | 20 mg LY3478045 (Part A) (N=6) | 60 mg LY3478045 (Part A) (N=6) | 180 mg LY3478045 (Part A) (N=6) | 500 mg LY3478045 (Part A) (N=6) | 700 mg LY3478045 (Part A) (N=6) | Placebo QD (Part B) (N=4) | Placebo QD + 40 mg Atorvastatin (Part B) (N=4) | 60 mg LY3478045 QD (Part B) (N=6) | 160 mg LY3478045 QD + 40 mg Atorvastatin (Part B) (N=6) | 300 mg LY3478045 QD (Part B) (N=6) | 360 mg LY3478045 QD + 40 mg Atorvastatin (Part B) (N=6)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT04270370/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT04270370/SAP_001.pdf